CLINICAL TRIAL: NCT01398774
Title: Altered Resting Energy Expenditure as a Cause of Obesity in Pseudohypoparathyroidism 1a: A Pilot Study
Brief Title: Energy Expenditure and Body Composition in Pseudohypoparathyroidism 1a
Status: Terminated | Type: Observational
Why Stopped: study expired
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 11-007972
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Pseudohypoparathyroidism Type 1A; Albright Hereditary Osteodystrophy
Keywords: Pseudohypoparathyroidism; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators would like to learn more about the metabolic consequences of pseudohypoparathyroidism type 1a in children, adolescents and adults with this condition. People with pseudohypoparathyroidism 1a are at risk for development of obesity. To better understand the cause of overweight or obesity, investigators are measuring body composition and resting energy expenditure (REE), which is the amount of calories burned while completely at rest. The investigators also want to determine the amount of body fat.

DETAILED DESCRIPTION:
Pseudohypoparathyroidism 1a (PHP1a) is a disorder that is associated with many endocrine problems. People with PHP1a are at risk for the development of obesity. The objective of the study will help determine if obesity is related to abnormalities energy expenditure, meaning that people with PHP1a may not burn as many calories while at rest as those without the disorder.

In order to further evaluate obesity in PHP1a, investigators are planning to measure resting energy expenditure (REE), which is the amount of calories burned while completely at rest. Investigators will also evaluate body composition by looking at measures of growth and development and determining the amount of body fat using dual energy x-ray absorptiometry (DXA) as well as blood and urine biologic markers of obesity. The investigators plan to evaluate people with PHP1a at all weights.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pseudohypoparathyroidism 1a
* Any body weight

Exclusion Criteria:

* Absence of above diagnosis

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects with Pseudohypoparathyroidism 1a
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2011-06; Primary Completion 2015-09 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 30 minutes
  The subject will rest for 30 minutes in the lab prior to the start of the test. A 60-minute resting energy expenditure (REE) test will be performed between 7:00 and 10:00 A.M. with the subject resting quietly under a clear, plastic hood watching a videotape.

SECONDARY OUTCOMES:
Characterize body composition in patients with PHP1a. | 12 months
  Body composition outcomes will be characterized by whole body lean mass and fat mass sex- and race-specific z-scores relative to height.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Levine, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Roizen JD, Danzig J, Groleau V, McCormack S, Casella A, Harrington J, Sochett E, Tershakovec A, Zemel BS, Stallings VA, Levine MA. Resting Energy Expenditure Is Decreased in Pseudohypoparathyroidism Type 1A. J Clin Endocrinol Metab. 2016 Mar;101(3):880-8. doi: 10.1210/jc.2015-3895. Epub 2015 Dec 28. PMID 26709970